CLINICAL TRIAL: NCT06619990
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study in Healthy Participants Followed by a Randomized, Double-Blind, Placebo-Controlled Phase 2 Study in Participants With Moderate-To-Severe Active Ulcerative Colitis.
Brief Title: Study of XmAb942 in Healthy Participants and Participants With Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XmAb942-01 (G942-101)
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Healthy Volunteers
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Active drug (Active Comparator): Active XmAb942 to be administered to healthy volunteers. Single administration of 3 ascending dose (SAD) levels of XmAb942 via SC (3 cohorts) or IV (3 cohorts) administration in 8 participants per cohort, randomized in a 3:1 ratio to active or placebo.
  Interventions: Biological: XmAb942
- Part A: Placebo (Placebo Comparator): Placebo Comparator to be administered to healthy volunteers. Single administration of 3 ascending dose (SAD) levels will be randomized in a 3:1 ratio to active or placebo.
  Interventions: Drug: Placebo
- Part B: Active (Active Comparator): Active XmAb942 to be administered to healthy volunteers. Multiple administrations of 2 ascending dose (MAD) levels of XmAb942 via IV administration in 8 participants per cohort, randomized in a 3:1 ratio to active or placebo.
  Interventions: Biological: XmAb942
- Part B: Placebo (Placebo Comparator): Placebo Comparator to be administered to healthy volunteers. Multiple administrations of 2 ascending dose (MAD) levels will be randomized in a 3:1 ratio to active or placebo.
  Interventions: Drug: Placebo
- Part C: Active (Active Comparator): Active XmAb942 to be administered to participants with moderately to severely active Ulcerative Colitis
  Interventions: Biological: XmAb942
- Part C: placebo (Placebo Comparator): Placebo comparator to be administered to participants with moderately to severely active Ulcerative Colitis
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: XmAb942 — Antibody
  Arms: Part A: Active drug; Part B: Active; Part C: Active
Drug: Placebo — Placebo
  Arms: Part A: Placebo; Part B: Placebo; Part C: placebo

SUMMARY:
Brief summary The Phase 1 study described herein will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of XmAb942 in healthy volunteers (Parts A and B). Part C of this study will be a Phase 2 study to evaluate XmAb942 in participants with ulcerative colitis (UC).

DETAILED DESCRIPTION:
This study consists of 3 parts, as follows:

Part A: Single ascending dose (SAD) in healthy participants, will entail administration of XmAb942 or matching placebo at 3 different dose levels of XmAb942.

Part B: Repeat dosing for up to 3 doses, will entail administration of XmAb942 or matching placebo at 2 different dose levels of XmAb942.

Part C: Participants with moderately to severely active UC to receive 3 different dose levels of XmAb942 or placebo during a 12-week induction period and single dose level of XmAb942 during a 40-week maintenance period, followed by a 24 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B

* Age 18-55
* Must be in good health with no significant medical history
* Clinical laboratory values within normal range
* BMI 18-35 (inclusive)
* Contraceptive use by men or women consistent with local regulations
* Able and willing to provide written informed consent

Part C

* Age 18-75
* Must be in good health with no significant medical history
* UC diagnosis ≥ 3 months prior to screening
* Diagnosis of moderately to severely active UC as defined by a (MMS) ≥ 5, with a MES ≥ 2 and RBS ≥ 1
* Evidence of UC extending ≥ 15 cm from the anal verge, as determined by screening colonoscopy
* Must have inadequate response to, loss of response to, or intolerance to at least 1 of the conventional or advanced therapies of UC
* Able and willing to provide written informed consent

Exclusion Criteria:

Parts A and B

* Any physical or psychological condition that prohibits study completion
* History of suicidal behavior or suicidal ideation
* Heavy use of nicotine containing products
* HIV, hepatitis B and hepatitis C positive
* Cardiac arrhythmia, or clinically significant abnormal ECG
* Active use of prescription medications within 14 days of Day -1
* Active use of over-the-counter, or herbal medication within 7 days of Screening
* Other investigational products within 30 days
* Blood or plasma donation within 60 days
* Pregnant or breastfeeding

Part C

* Any physical or psychological condition that prohibits study participation
* Diagnosis of Crohn disease, indeterminate colitis, indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, and diverticular disease associated with colitis.
* Positive screen for Clostridium difficile (C. Difficile) toxins
* HIV, hepatitis B and hepatitis C positive
* Cardiac arrhythmia, or clinically significant abnormal ECG
* Pregnant or breastfeeding

Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of XmAb942 in healthy volunteers (Part A) | 20 weeks
Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of XmAb942 in healthy volunteers (Part B) | 28 weeks
Clinical remission based on modified mayo score (MMS), defined as MMS ≤ 2 with Mayo endoscopic score (MES) of 1, rectal bleeding subscore (RBS) of 0, and stool frequency subscore (SFS) of 0-1. | 12 weeks
  A composite score of ulcerative colitis (UC) disease activity on a scale of increasing severity from 0-9. It is calculated by adding the results from Mayo endoscopic subscore (MES) which measures GI bleeding, stool frequency subscore (SFS) which measures stool frequency per day, and rectal bleeding subscore (RBS), which measures presence of blood during stool passing. Each subscore is a scale of increasing severity from 0 to 3.

SECONDARY OUTCOMES:
Serum PK parameters of XmAb942 in Healthy Volunteers (Part A) | up to 20 weeks
  • Cmax (Maximum concentration of drug)
Serum PK parameters of XmAb942 in Healthy Volunteers (Part A) | up to 20 weeks
  • AUC0-last (Area under the curve drug concentration-time curve to last concentration)
Serum PK parameters of XmAb942 in Healthy Volunteers (Part B) | up to 28 weeks
  • Cmax (Maximum concentration of drug)
Serum PK parameters of XmAb942 in Healthy Volunteers (Part B) | up to 28 weeks
  • AUC0-tau AUC within a dosing interval, calculated using the linear trapezoidal rule
Incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) (Part C) | 72 weeks
Discontinuations due to TEAEs (Part C) | 72 weeks
Endoscopic improvement defined as (MES) of 0 or 1 (Part C). | 12 weeks
Change from baseline in MS (Part C). | 12 weeks
Clinical response based on MMS score (Part C) defined as decrease from baseline in the MMS of ≥ 2 points and at least a 30% reduction from baseline, and decrease of ≥ 1 point in RBS from baseline or absolute RBS ≤ 1 | 12 weeks
Histological improvement as determined by change in Robarts Histopathology Index (RHI) scores, ranging from 0 (no disease activity) to 33 (severe disease activity). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Osterman, MD, MSCE, Study Director — Xencor, Inc.
Locations (20):
- United States (7):
  - Xencor Investigative Site, Scottsdale, Arizona
  - Xencpr Investigative Site, Jacksonville, Florida
  - Xencor Investigative Site, Kissimmee, Florida
  - Xencor Investigative Site, Tampa, Florida
  - Xencor Investigative Site, Raleigh, North Carolina
  - Xencor Investigative Site, Kingwood, Texas
  - Xencor Investigative Site, San Antonio, Texas
- Australia (4):
  - Xencor Investigative Site, Wollongong, New South Wales
  - Xencor Investigative Site, South Brisbane, Queensland
  - Xencor Investigative Site, Joondalup, Western Australia
  - Xencor Investigative Site, Nedlands, Western Australia
- Xencor Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Xencor Investigative Site, London, Ontario
  - Xencor Investigative Site, Scarborough Village, Ontario
- Xencor Investigative Site, Tbilisi, Georgia
- Xencor Investigative Site, Chisinau, Moldova
- Xencor Investigative Site, Szczecin, Poland
- Ukraine (3):
  - Xencor Investigative Site, Ivano-Frankivsk
  - Xencor Investigative Site, Kyiv
  - Xencor Investigative Site, Lviv

IPD SHARING:
Plan to Share IPD: No